CLINICAL TRIAL: NCT07149675
Title: A Multi-center Prospective-retrospective Study of the Clinical Characteristics, Biochemical Response, and Long-term Outcomes in Patients With Primary Biliary Cholangitis
Brief Title: PBC Long-term Outcomes Study
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jidong Jia, Principal Investigator, Beijing Friendship Hospital
Other Study IDs: 2025-P2-173-01
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Primary Biliary Cholangitis (PBC); Long-term Outcomes; Prognosis; Multicenter Prospective Study
Keywords: Primary biliary cholangitis; long-term outcomes; prognosis; multicenter; Symptoms
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PBC cohort: PBC Cohort from multicenters across multiple provinces and cities nationwide in China

SUMMARY:
Primary biliary cholangitis (PBC) is an autoimmune liver disease predominantly affecting middle-aged women. While historically it was deemed rare, advancements in specific auto-antibody tests have led to increased recognition of PBC. The long-term survival of PBC patients in China is not yet fully understood. Several studies have investigated the prognosis of PBC in China. While these studies provide valuable insights into the disease characteristics and prognostic factors of PBC in China, they are all single-center studies with limitations. They lack consideration of the impact of symptoms, varying disease stages, and second-line treatments on prognosis. Therefore, there is a pressing need for multicenter and large-scale studies to further elucidate the characteristics and long-term survival of PBC patients in China.

Biochemical response to ursodeoxycholic acid (UDCA) is an independent factor associated with long-term survival. Unfortunately, approximately 30-40% of PBC patients demonstrate insufficient biochemical response to UDCA. In our cohort, we reported a higher nonresponse rate, with about 44% according to the Paris I criteria. These patients remain at risk for disease progression to advanced stages and may benefit from additional second-line drug therapies. With significant advancements in the development of new drugs for PBC, a comprehensive understanding of patients with suboptimal responses to UDCA-including long-term prognosis, the distribution of different disease stages, and the prevalence of pruritus-will provide a basis for individualized treatment strategies.

Additionally, fatigue and pruritus are prevalent symptoms for PBC patients and fluctuates independently of disease activity or stage, which significantly diminishing health-related quality of life. However, the incidence and impact of fatigue and pruritus on long-term outcomes for PBC patients in China need further clarification.

Therefore, we would like to conduct this multicenter study to estimate the prevalence of PBC in China and to evaluate the symptomatic burden, treatment, and long-term outcomes among PBC patients in China.

DETAILED DESCRIPTION:
This is a retrospective-prospective, multicenter cohort study that plans to enroll approximately 4,000 patients with PBC from ten centers across multiple provinces and cities nationwide of China.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis consistent with PBC.
* Willingness to participate, with informed consent obtained from the patient or legal representative (if the patient is deceased or cognitively impaired), and ability to adhere to follow-up.

Exclusion Criteria:

* Co-existing chronic hepatitis B or C, drug-induced liver injury, autoimmune hepatitis, primary sclerosing cholangitis, or hereditary/metabolic liver diseases.
* Co-existingMalignancy or severe cardiac, pulmonary, renal, cerebral, or hematologic disorders expected to substantially shorten life expectancy.
* Incomplete baseline medical records or laboratory data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PBC patients from ten centers across multiple provinces and cities nationwide of China.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-05-18 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
death and/or liver transplantation. | From January 2000 to December 2029

SECONDARY OUTCOMES:
Liver-related adverse events | From January 2000 to December 2025
  ascites, esophageal-gastric variceal bleeding, hepatic encephalopathy, hepatocellular carcinoma, liver failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Research Center, Beijing Friendship Hospital, Capital Medical University, Beijing, Select A State Or Province, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen S, Li MQ, Duan WJ, Li BE, Li SX, Lv TT, Ma L, Jia JD. Concomitant extrahepatic autoimmune diseases do not compromise the long-term outcomes of primary biliary cholangitis. Hepatobiliary Pancreat Dis Int. 2022 Dec;21(6):577-582. doi: 10.1016/j.hbpd.2022.05.009. Epub 2022 May 24. PMID 35668014
- [Background] Zeng N, Duan W, Chen S, Wu S, Ma H, Ou X, You H, Kong Y, Jia J. Epidemiology and clinical course of primary biliary cholangitis in the Asia-Pacific region: a systematic review and meta-analysis. Hepatol Int. 2019 Nov;13(6):788-799. doi: 10.1007/s12072-019-09984-x. Epub 2019 Sep 25. PMID 31552558
- [Background] You H, Ma X, Efe C, Wang G, Jeong SH, Abe K, Duan W, Chen S, Kong Y, Zhang D, Wei L, Wang FS, Lin HC, Yang JM, Tanwandee T, Gani RA, Payawal DA, Sharma BC, Hou J, Yokosuka O, Dokmeci AK, Crawford D, Kao JH, Piratvisuth T, Suh DJ, Lesmana LA, Sollano J, Lau G, Sarin SK, Omata M, Tanaka A, Jia J. APASL clinical practice guidance: the diagnosis and management of patients with primary biliary cholangitis. Hepatol Int. 2022 Feb;16(1):1-23. doi: 10.1007/s12072-021-10276-6. Epub 2022 Feb 4. No abstract available. PMID 35119627